CLINICAL TRIAL: NCT01452503
Title: Assessing Preference for 3 Female Condoms: A Comparative Evaluation of the PATH Woman's Condom, FC2 and the Reddy 6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 9928; USAID (Other Grant/Funding Number: GPO-A-00-05-00022-00;(W0118))
Record Dates: First submitted 2011-08-19; First posted 2011-10-17 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Contraception
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonization; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PATH Women's Condom (Active Comparator): PATH Women's Condom
  Interventions: Device: Path Women's Condom
- FC2 female condom (Active Comparator): Female Health Company's FC2 female condom
  Interventions: Device: FC2 female condom
- Reddy 6 female condom (V-Amour) (Active Comparator): Reddy 6 female condom (Commercially known as the V-Amour female condom)
  Interventions: Device: Reddy 6 female condom (V-Amour)

INTERVENTIONS:
Device: Path Women's Condom — comparison between 3 types of female condoms
  Arms: PATH Women's Condom
Device: FC2 female condom — comparison between 3 types of female condoms
  Arms: FC2 female condom
Device: Reddy 6 female condom (V-Amour) — comparison between 3 types of female condoms
  Arms: Reddy 6 female condom (V-Amour)

SUMMARY:
Evaluation of preference for three female condoms (FC).

DETAILED DESCRIPTION:
The primary goal of this study was to identify the female condom most preferred by study participants. This provided USAID with data to make informed decisions regarding female condom purchases. The study was conducted in three parts. The objective of Part 1 was to familiarize each participant with the three FC types, to minimize learning curve effect in subsequent phases of study, and to gather information on participant demographics, FC acceptability, device function, safety, preference for each of the condom types, and use of male condoms during the same time period. The objective of Part 2 was to determine actual, "unstated" and "unbiased" preference for a particular type of FC. The objective of Part 3 was to identify reasons for preference of a particular FC type and to document details surrounding product use/non-use.

ELIGIBILITY:
Inclusion Criteria:

* All women enrolled in this research must meet the following selection criteria:

  1. must be at least 18 years of age.
  2. must be literate (able to read a newspaper or letter easily).
  3. must be sexually active (defined as having at least two vaginal coital acts per week and not being abstinent in the month prior to enrollment).
  4. must be in an exclusive (monogamous) sexual relationship with her spouse or partner while participating in this research study.
  5. must have been in a sexual relationship with this partner for at least 6 months.
  6. must be without evidence of STI as determined through syndromic diagnosis and vaginal examination.
  7. must be on hormonal or other non-barrier contraception (e.g. OCs, injectables, IUD, or have had a tubal sterilization or be post-menopausal-defined as 12 months with no period).
  8. must be willing to give informed consent.
  9. must be able to complete condom use log.
  10. must be willing to use the study condoms as directed.
  11. must be willing to adhere to the follow-up schedule and all study procedures.
  12. must have successfully completed a given phase of study before advancing into subsequent phases (e.g. successfully completing Part 1 before advancing to Part 2, etc.).
  13. must be willing to provide research study staff with an address, phone number or other locator information while participating in the study.
  14. must be willing to participate in the study for up to six months.
* Exclusion Criteria:

  1. must not be a sex worker.
  2. must not be pregnant (as determined by pregnancy testing) or planning a pregnancy during the time of the research study.
  3. must not be breastfeeding.
  4. must not have known sensitivities or allergies to latex, polyurethane, vaginal/sexual lubricants or the lubricants used on condoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Preference of female condom by type | 3 months
  The objective of Part 1 is to familiarize each participant with the use characteristics of the three female condom types in order to minimize learning curve effect in subsequent phases of study. In Part 2, a 'simulated market' will be created in order to determine an unbiased, free choice preference for a particular FC type. Part 3 will detail the reasons for participants' selection/preference of specific FC types.

SECONDARY OUTCOMES:
Safety of each of the female condom types | 3 months
  safety measured by number of particpants with adverse events
Function of each of the female condom types | 3 Months
  FC function measured by number of female condoms that failed during use (e.g. breakage, slippage and invagination) as self-reported by subjects through coital logs

CONTACTS AND LOCATIONS:
Overall Officials: Mags Beksinska, MSc. PhD, Principal Investigator — RHRU
Locations (1):
- Commercial City Clinic Department of Health, Durban, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beksinska M, Smit J, Joanis C, Hart C. Practice makes perfect: reduction in female condom failures and user problems with short-term experience in a randomized trial. Contraception. 2012 Aug;86(2):127-31. doi: 10.1016/j.contraception.2011.11.071. Epub 2012 Jan 20. PMID 22264667